CLINICAL TRIAL: NCT07049588
Title: A Multi-omic Approach to the Identification of Novel Biomarkers in Early Charcot-Marie-Tooth 1A Disease (CMT1A)
Brief Title: Identification of Novel Biomarkers in Early Charcot-Marie-Tooth 1A Disease
Acronym: CMT-MODS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other); University Medical Center Göttingen (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RCAPHM24_0381; 2024-A02403-44 (Other: ID RCB)
Record Dates: First submitted 2025-06-13; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Charcot-Marie-Tooth Disease Type 1A
Keywords: CMT1A; Fat Fraction; CMT Examination Score Rasch; CMT Functional Outcome Measure; Skin Biopsy; histological markers; MRI muscle
MeSH Terms: conditions — Charcot-Marie-Tooth Disease | interventions — Hematologic Tests

STUDY DESIGN:
Intervention Model Description: Comparison of patient and healthy volunteers data at inclusion (M0) and 12 months (M12)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Charcot-Marie-Tooth Neuropathy 1A (Other): Patient with genetically confirmed CMT1A or with a parent whose diagnosis is genetically confirmed,
  Interventions: Other: Quantitative neuromuscular MRI; Other: Skin biopsy; Other: Clinical scores; Other: Blood test; Other: Patient Report Outcomes Measures
- Healthy volunteers (Other): Patient-matched controls
  Interventions: Other: Quantitative neuromuscular MRI; Other: Skin biopsy; Other: Clinical scores; Other: Blood test

INTERVENTIONS:
Other: Quantitative neuromuscular MRI — Quantification of biomarkers as fat fraction, magnetization Transfer Ratio, muscular volume, relaxation time T2
Other: Skin biopsy — Performed on the arm or index finger, depending on patient age
Other: Clinical scores — ONLS, CMTES-R, CMT-Peds, CMT-FOM
Other: Blood test — 10 ml sample
Other: Patient Report Outcomes Measures — pCMT-QoL, EVA, WALK-12, PGI-c, SF-12
  Arms: Charcot-Marie-Tooth Neuropathy 1A

SUMMARY:
This is a 2-year follow-up study of a cohort of 35 CMT1A patients and 20 healthy volunteers. The main objective is identifying prognostic markers for CMT1A using multi-omics analysis. The study is recruiting subjects between the ages of 10 and 30.

The most common inherited neuropathy is Charcot-Marie-Tooth disease type 1A (CMT1A), caused by a duplication of the gene expressing PMP22. CMT1A patients develop symptoms in early childhood with variable progression and there is no established therapy until now. Therapy must start in childhood, before peripheral nerves degenerate. However, we lack easily obtainable biomarkers in early disease stages.

In CMT-MODs, we will identify disease and prognostic biomarkers in young CMT1A patients.

DETAILED DESCRIPTION:
The CMT-MODs project aims to conduct a multi-omics analysis (transcriptomics, proteomics, lipidomics) in young patients with early-stage CMT1A. This evaluation should enable the identification of prognostic and change-sensitive biomarkers for use in clinical trials.

A large cohort of CMT1A children, adolescents and young adults aged 10-30 years over 12 months applying the novel clinical outcome measures CMT Examination Score/CMT Neuropathy Score Version Version 2 Rasch versions (CMTES-R/CMTNSv2-R), the functional outcome measure CMT-FOM, pCMT-Qol, as well as a nerve conduction study (NCS) and quantitative MRI will be assessed.

Blood (and optional skin) samples will be taken and gene expression of the most promising candidates will be identified.

This assessment of CMT patients at early disease stages will allow CMT-MODs to establish biomarkers that may serve as a standard readout for disease severity and predict the disease course.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer or patient who has given consent for participation in the study or, for minors, a healthy volunteer whose two parents have given consent for participation in the study.
* Patient with genetically confirmed CMT1A or with a parent whose diagnosis is genetically confirmed
* Patient able to walk with or without assistance

Exclusion Criteria:

* Healthy volunteer with neurological disorders
* Healthy volunteer or patient with a contraindication to MRI,
* Healthy volunteers or patient under 30 kg
* Helathy volunteer on long-term therapy
* Patient with other neuromuscular pathologies
* Patient in a period of exclusion from another research protocol at the time of signing the consent/non-opposition form
* Pregnant or breast-feeding women
* Subjects covered by articles L1121-5 to 1121-8 of the French Public Health Code (minors, adults under guardianship or trusteeship, patients deprived of their liberty, pregnant or breast-feeding women)
* Subjects who cannot read and understand the French language well enough to be able to give their consent to participate in research

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-06-24 (Estimated); Primary Completion 2027-06-24 (Estimated); Study Completion 2028-06-24 (Estimated)

PRIMARY OUTCOMES:
Transcriptomic analysis | Between inclusion (month 0) and one year later (month 12)
  RNA seq on blood and skin tissues
Proteomic analysis | Between inclusion (month 0) and one year later (month 12)
  Label-free quantitative approach on blood and skin tissues

SECONDARY OUTCOMES:
MRI muscle biomarkers : Fat Fraction measure | Between inclusion (month 0) and one year later (month12)
MRI muscle biomarkers : Magnetization Transfer Ratio | Between inclusion (month 0) and one year later (month12)
MRI muscle biomarkers : T2 relaxation time | Between inclusion (month 0) and one year later (month12)
MRI muscle biomarkers : muscle volume | Between inclusion (month 0) and one year later (month12)
Clinical score : ONLS | Between inclusion (month 0) and one year later (month12)
  Overall Neuropathy Limitations Scale
Clinical score : CMTES-R | Between inclusion (month 0) and one year later (month12)
  CMT Examination Score
Clinical score : CMT-FOM | Between inclusion (month 0) and one year later (month12)
  The CMT-Functional Outcome Measure
Clinical score : CMT-Peds | Between inclusion (month 0) and one year later (month 12)
  Charcot-Marie-Tooth Disease Pediatric Scale
PROM (Patient Reported Outcomes Measures) : pCMT-QoL | Between inclusion (month 0), month 6, and one year later (month12)
  Pediatrics CMT Questionnaire of Life
PROM (Patient Reported Outcomes Measures) : VAS | Between inclusion (month 0), month 6, and one year later (month 12)
  Visual Analog Scale
PROM (Patient Reported Outcomes Measures) : WALK-12 | Between inclusion (month 0), month 6, and one year later (month 12)
PROM (Patient Reported Outcomes Measures) : PGI-c | Between inclusion (month), month 6, and one year later (month 12)
  Patient's Global Impression of change scale
PROM (Patient Reported Outcomes Measures) : SF-12 | Between inclusion (month 0), month 6, and one year later (month12)

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — Assistance Publique - Hôpitaux de Marseille
Locations (1):
- Assistance Publique - Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No